CLINICAL TRIAL: NCT03274011
Title: Efficacy and Safety of Apatinib for Recurrent or Metastatic Esophageal Squamous Cell Carcinoma: A Phase II, Prospective, Single-arm, Multicenter Trial
Brief Title: Efficacy and Safety of Apatinib for Recurrent or Metastatic Esophageal Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Kuai Le Zhao, MD, Chief of Chest Radiation Oncology Department, Fudan University Cancer Center, Shanghai, P.R. China, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESO-Shanghai11
Record Dates: First submitted 2017-08-20; First posted 2017-09-06 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2019-02

CONDITIONS: Esophageal Neoplasms
MeSH Terms: conditions — Esophageal Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib Treatment (Experimental): Apatinib for Recurrent or Metastatic Esophageal Squamous Cell Carcinoma
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Apatinib is a small-molecule tyrosine kinase inhibitor (TKI) that highly selectively binds to and strongly inhibits vascular en-dothelial growth factor receptor 2 (VEGFR-2), with a decrease in VEGF-mediated endothelial cell migration, proliferation, and tumor microvascular density. Previous data showed that apatinib treatment significantly improved OS and PFS with an acceptable safety profile in patients with advanced gastric cancer refractory to two or more lines of prior chemotherapy. Our study will observe the efficacy and safety of Apatinib for recurrent or metastatic esophageal squamous cell carcinoma: A phase II, prospective, single-arm, multicenter trial.

SUMMARY:
There is no standard treatment strategy for recurrent or metastatic esophageal squamous cell carcinoma patients now, especially after the second-line treatment. Most of the patients have the bad ECOG (Eastern Cooperative Oncology Group) score and prognosis. Chemotherapy, radiotherapy, surgery are usually unacceptable for them. Previous data showed that apatinib treatment significantly improved OS(overall survival) and PFS(progression-free survival) with an acceptable safety profile in patients with advanced gastric cancer refractory to two or more lines of prior chemotherapy. The study will observe the efficacy and safety of Apatinib for recurrent or metastatic esophageal squamous cell carcinoma: A phase II, prospective, single-arm, multicenter trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age: ≥18 years old
2. An ECOG score of 0-2
3. Pathologically diagnosed with Esophageal Squamous Cell Carcinoma.
4. At least second-line treatment failure regimens without targeted therapy.
5. Measurable lesion.
6. An expected survival of ≥ 3 months.
7. Major organ function had to meet the following criteria:

1)For regular test results: HB(hemoglobin) ≥ 90g / L (14 days without blood transfusion); ANC(absolute neutrophil count) ≥ 1.5 × 109 / L; PLT(platelet) ≥ 80 × 109 / L 2)Biochemical tests results: Bilirubin <1.5 times the upper limit of normal (ULN) ALT(Alanine aminotransferase) and AST≤2.5 × ULN; liver metastases, if any, the ALT and AST≤5 × ULN; Endogenous creatinine clearance≥50ml/min (Cockcroft-Gault formula) 8. Informing consent.

Exclusion Criteria:

1. Previously or presently suffering from other malignancies, except for the cured and stable carcinoma;
2. Pregnant or lactating women;
3. Participation in clinical trials with other drugs in the preceding four weeks.
4. Factors that could have an effect on oral medication (such as inability to swallow, chronic diarrhea and intestinal obstruction).
5. Serious bleeding events within 4weeks (≥3 degree)-CTCAE(Common Terminology Criteria for Adverse Events) 4.0
6. Central nervous system metastasis or a history of central nervous system metastasis.
7. Hypertension and antihypertensive drug treatment that does not normalize blood pressures (systolic blood pressure> 140 mmHg and diastolic blood pressure > 90 mm Hg); With unstable angina pectoris; Arrhythmia; Coronary heart disease greater than Class II; Angina pectoris diagnosed with 3 months or myocardial infarction event occurs within 6 months before recruiting.
8. With the open wounds or fractura.
9. A history of organ transplant.
10. Coagulation dysfunction (PT(prothrombin time)>16 s, APTT(activated partial thromboplastin time)>43 s, TT(thrombin time)>21 s, Fbg(Fibrinogen)<2g/L), a tendency to bleed or receiving thrombolytic or anticoagulant therapy.
11. A history of abuse of psychotropic drugs or mental disorders.
12. Central nervous system disorders.
13. A history of immunodeficiency.
14. Arterial/venous thrombosis events within 12 months before recruiting.
15. Use of CFDA(China Food and Drug Administration) approved anti-gastric modern traditional Chinese medicine preparations and immunomodulatory agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 12 weeks
  the time with no progression from the treatment

SECONDARY OUTCOMES:
Overall Survival | 24 weeks
  the time from the treatment to death
Overall Response Rate | 4 weeks
  partial response and complete response

CONTACTS AND LOCATIONS:
Overall Officials: kuaile zhao, doctor, Principal Investigator — Radiation Oncology Department, Fudan University Cancer Center, Shanghai, P.R. China.
Locations (1):
- Shanghai Yangpu District East Hospital, Shanghai, Shanghai Municipality, China